CLINICAL TRIAL: NCT04748835
Title: Investigating Factors Related to Nutritional Intake and Weight Gain Among Those With SCI Over the First 12 Months Following Discharge From Inpatient Rehabilitation
Brief Title: The SEEA (SCI Energy Expenditure and Activity) Study
Acronym: SEEA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Baylor Research Institute (Other)
Responsible Party: Principal Investigator, Katherine Froehlich-Grobe, Director of Rehabilitation Research, Baylor Research Institute
Other Study IDs: 016-277
Record Dates: First submitted 2020-10-22; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Spinal Cord Injuries; Obesity; Metabolic Syndrome; Cardiovascular Diseases; Diet Habit
MeSH Terms: conditions — Spinal Cord Injuries; Obesity; Metabolic Syndrome; Cardiovascular Diseases; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
People with SCI are at higher risk of obesity and chronic diseases, such as hypertension, high cholesterol, diabetes and cardiovascular disease, than the general population. Researchers currently lack data on factors that influence weight gain among people with SCI. During this one-year observational study, study staff will enroll 60 individuals with SCI while they are inpatients at Baylor Scott & White Institute for Rehabilitation (BSWIR). Data will be collected at 3 time periods (before discharge and 6 and 12 months after discharge) in order to better understand factors that affect weight gain over the first 12 months following discharge from inpatient rehabilitation, such as nutritional intake, environmental access, psychosocial factors, energy requirements and risk factors for metabolic syndrome. These data will be used to inform future interventions for people with SCI.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years with complete or incomplete spinal cord injury (SCI)
* Currently have or are expected to regain enough arm function within 6 months to feed themselves independently.
* Injury occurred within previous 18 months

Exclusion Criteria:

* Unwilling or unable to complete repeat assessments
* Cognitive impairment or brain injury that limits ability to provide data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study participants are people who have incurred a spinal cord injury within the previous 18 months prior to study enrollment who have been admitted to inpatient rehabilitation at Baylor Scott & White Institute for Rehabilitation in Dallas, TX. Participants must have or be expected to regain enough arm/hand function to feed themselves independently and be willing and able to complete physical measurements and surveys.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in nutritional intake | 1 year
  Measure self-report and hospital reported average daily caloric intake, macronutrients (protein, fats, carbohydrates), and micronutrient (sodium) over 3 days at each study time point: baseline, 6 months, and 1 year
Changes in environmental access to kitchen appliances and self-reported limitations and assistance needed for selecting, preparing, and eating meals. | 1 year
  Using the Assessment of life habits survey (abbreviated as LIFE-H) to determine the proportion of individuals with SCI who require assistance using kitchen appliances and preparing meals. Additional qualitative analyses will include examining the digital photos for intra-individual variation across time to determine whether there are changes to improve access to kitchen spaces and appliances.
Correlation between psychosocial factors (mood, stress, coping, and sleep) and caloric intake | 1 year
  Mood will be measured using the Positive and Negative Affect States Scale (PANAS); stress will be measured using the Perceived Stress Scale (PSS-4); coping will be measuring using the Daily Coping Inventory (DCI); sleep will be measured with the Pittsburgh Sleep Quality Index (PSQI). Caloric intake is measured through participant self-report through the HealthWatch 360 app, the Automated Self-Administered Recall System (ASA-24) or through hospital records.
Changes in resting metabolic rate | 1 year
  As measured by resting metabolic rate using a MedGem device
Time spent performing physical activity | 1 year
  Time spent performing physical activity at each of the study timepoints will be measured using an Actigraph device

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Froehlich-Grobe, PhD, Principal Investigator — Baylor Scott & White Institute for Rehabilitation
Locations (1):
- Baylor Scott & White Institute for Rehabilitation - Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided